CLINICAL TRIAL: NCT01096589
Title: Preliminary Study to Assess the Effectiveness of 3M Oedema Reduction System in the Treatment of Lymphoedema Treatment Compared to Comprilan Short-stretch Bandage Compression Therapy
Brief Title: Assessment of 3M Oedema Reduction System in the Treatment of Lymphoedema Compared to Commercial Short-stretch Bandage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU Study-05-000012
Record Dates: First submitted 2010-03-22; First posted 2010-03-31 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Lymphedema
Keywords: lymphoedema; lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 - 3M Coban 2 (Experimental): 3M Coban 2 - 2 apps/wk
  Interventions: Device: 3M Coban 2 (Compression System)
- Arm 2 - 3M Coban 2 (Experimental): 3M Coban 2 - 3 apps/wk
  Interventions: Device: 3M Coban 2 (Compression System)
- Arm 3 - 3M Coban 2 (Experimental): Arm 3 - 3M Coban 2 - 5 apps/wk
  Interventions: Device: 3M Coban 2 (Compression System)
- Arm 4 - Comprilan (Active Comparator): Comprilan short-stretch bandage 5 apps/wk
  Interventions: Device: Comprilan

INTERVENTIONS:
Device: 3M Coban 2 (Compression System) — Nonwoven cohesive backing and foam.
  Arms: Arm 1 - 3M Coban 2
Device: 3M Coban 2 (Compression System) — Nonwoven cohesive backing and foam.
  Arms: Arm 2 - 3M Coban 2
Device: 3M Coban 2 (Compression System) — Nonwoven cohesive backing and foam.
  Arms: Arm 3 - 3M Coban 2
Device: Comprilan — Commercial short-stretch bandage (Comprilan; BSN Medical Ltd, Hull, U.K).
  Arms: Arm 4 - Comprilan

SUMMARY:
Objectives. The primary objective of the study is to assess volume reduction in the treatment of lymphoedematous legs and arms with compression bandaging.

Secondary objectives:

* Assessment of safety
* Quality of life
* Health economic parameters
* Slippage
* Subbandage pressure

ELIGIBILITY:
Inclusion Criteria (Arm):

* Mobile males or females, age 18 years or older
* Unilateral arm lymphoedema of secondary origin
* Pitting arm lymphoedema diagnosed as stage II or late stage II according to the International Society of Lymphology staging
* Patients who require intense bandaging therapy (approx. >= 15% increase in arm volume over the opposite healthy arm)
* Completion of all primary and adjuvant cancer treatments (surgery, chemotherapy, radiotherapy) at least 6 months prior to randomisation
* Willing to give written informed consent and willing to comply with the study protocol

Inclusion Criteria (Leg):

* Mobile males or females, age 18 years or older
* Unilateral or bilateral leg lymphoedema of primary or secondary origin
* Pitting leg lymphoedema diagnosed as stage II or late stage II according to the International Society of Lymphology staging
* Patients who require intense bandaging therapy
* Completion of all primary and adjuvant cancer treatments (surgery, chemotherapy, radiotherapy) at least 6 months prior to randomisation
* Willing to give written informed consent and willing to comply with the study protocol

Exclusion Criteria (Arm):

* Known pregnancy
* Evidence of active cancer, either local or metastatic
* A period of intense daily bandaging within the last month
* Decompensated heart failure or clinically relevant kidney or liver disease
* Known relevant arterial disease of the arms
* Deep vein thrombosis or phlebitis in the last 3 months
* Paralysis of the arms
* Clinical infection of the arms (e.g. erysipelas)
* Wounds located at the study arm that require dressing change more than once a week
* History of allergic reactions to study material
* Participation in any prospective clinical study that can potentially interfere with this study
* Participants who are, in the opinion of the clinical investigator, unsuitable for enrolment in this study, for reasons not specified in the exclusion criteria.

Exclusion Criteria (Leg):

* Known pregnancy
* Evidence of active cancer, either local or metastatic
* A period of intense daily bandaging within the last month
* Decompensated heart failure or clinically relevant kidney or liver disease
* Deep vein thrombosis or phlebitis in the last 3 months
* Known relevant arterial disease of the legs
* Paralysis of the legs
* Clinical infection of the legs (e.g. erysipelas)
* Circumferential Lymphorrhoea
* Wounds located at the study leg that require dressing change more than once a week
* History of allergic reactions to study material
* Participation in any prospective clinical study that can potentially interfere with this study
* Participants who are, in the opinion of the clinical investigator, unsuitable for enrolment in this study, for reasons not specified in the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Moffatt, Prof., Principal Investigator — Faculty of Medicine, Division of Nursing and Healthcare, Universtity of Glasgow, G12 8LW
Locations (11):
- United States (4):
  - NorthShore University Healthsystem, Evanston, Illinois
  - University of Missouri, Columbia, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Memorial Hermann Hyperbaric Center, Houston, Texas
- United Kingdom (7):
  - 56 London Road Clinic, Milborne Port, Dorset
  - Kendal Lymphology Centre, Kendal
  - LOROS Hospice, Leicester
  - St Giles Hospice Lymphoedema Service, Lichfield
  - Enfield Macmillan Lymphoedema Service, London
  - St Oswalds Hospice Lymphoedema Clinic, Newcastle upon Tyne
  - Swansea Lymphoedema Service Singleton Hospital, Swansea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomly allocated to the 4 application frequencies for 19 days.
  The randomisation was stratified according to limb location. Enroled participants were randomly assigned to one of the four treatment groups. Patients were treated in private lymphoedema clinics or in NHS centres (UK). US patients were treated in hospitals.
Groups:
- Arm 1 - 3M Oedema Reduction System: 3M Oedema Reduction System - 2 apps/wk
  3M Oedema Reduction System (Compression Bandage) : Nonwoven cohesive backing and foam.
- Arm 2 - 3M Oedema Reduction System: 3M Oedema Reduction System - 3 apps/wk
  3M Oedema Reduction System (Compression Bandage) : Nonwoven cohesive backing and foam.
- Arm 3 - 3M Oedema Reduction System: 3M Oedema Reduction System - 5 apps/wk
  3M Oedema Reduction System (Compression Bandage) : Nonwoven cohesive backing and foam.
- Arm 4 - Commercial Compression System 5 Apps/wk: Commercial Compression System 5 apps/wk
  Short-stretch Bandage (Comprilan; BSN Medical Ltd,). : Commercial short-stretch bandage (Comprilan; BSN Medical Ltd, Hull, U.K).
Period: Overall Study
Arm/Group | Arm 1 - 3M Oedema Reduction System | Arm 2 - 3M Oedema Reduction System | Arm 3 - 3M Oedema Reduction System | Arm 4 - Commercial Compression System 5 Apps/wk
Started | 22 | 20 | 22 | 18
Completed | 18 | 18 | 18 | 15
Not Completed | 4 | 2 | 4 | 3
Not completed — Adverse Event | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1
Not completed — Compliance with protocol | 0 | 0 | 1 | 0
Not completed — found treatment exhausting | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - 3M Oedema Reduction System | Arm 2 - 3M Oedema Reduction System | Arm 3 - 3M Oedema Reduction System | Arm 4 - Commercial Compression System 5 Apps/wk | Total
Number analyzed (Participants) | 22 | 20 | 22 | 18 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 11 | 14 | 49
  >=65 years | 7 | 11 | 11 | 4 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.73 (13.29) | 61.85 (14.49) | 62.27 (13.25) | 56.22 (14.78) | 60.16 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 17 | 77
  Male | 2 | 0 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 2 | 2 | 12
  United Kingdom | 17 | 17 | 20 | 16 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percent Volume Change of Affected Limb at End of Treatment Compared to Baseline.
Time Frame: baseline and after 3 weeks of treatment
Population: Patients must have completed the first week.
Measure: Mean (Standard Deviation); unit: % volume change measured in mL.
Arm/Group | Arm 1 - 3M Oedema Reduction System | Arm 2 - 3M Oedema Reduction System | Arm 3 - 3M Oedema Reduction System | Arm 4 - Commercial Compression System 5 Apps/wk
Number analyzed (Participants) | 18 | 20 | 22 | 16
% volume change measured in mL. | -14.56 (12.22) | -7.09 (7.30) | -10.24 (8.65) | -9.84 (4.34)

2. Secondary Outcome: Assessment of Safety by Incidence of Adverse Events.
Time Frame: 3 weeks
Measure: Number; unit: No. of treatment-emergent adverse events
Arm/Group | Arm 1 - 3M Coban 2 | Arm 2 - 3M Coban 2 | Arm 3 - 3M Coban 2 | Arm 4 - Comprilan
Number analyzed (Participants) | 22 | 20 | 22 | 18
No. of treatment-emergent adverse events | 13 | 11 | 14 | 10

ADVERSE EVENTS:
Arm/Group | Arm 1 - 3M Oedema Reduction System | Arm 2 - 3M Oedema Reduction System | Arm 3 - 3M Oedema Reduction System | Arm 4 - Commercial Compression System 5 Apps/wk
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 13/22 | 11/20 | 14/22 | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - 3M Oedema Reduction System (N=22) | Arm 2 - 3M Oedema Reduction System (N=20) | Arm 3 - 3M Oedema Reduction System (N=22) | Arm 4 - Commercial Compression System 5 Apps/wk (N=18)
Medical device discomfort (General disorders) | 2 (2) | 3 (5) | 2 (4) | 3 (6)
Application site discomfort (General disorders) | 0 (0) | 1 (1) | 4 (5) | 2 (3)
Application site irritation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site paraethesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (3) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site vesicles (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less